CLINICAL TRIAL: NCT00497081
Title: Mirtazapine to Reduce Methamphetamine Use Among MSM With High-risk HIV Behaviors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: San Francisco Department of Public Health (Other Government)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Public Health Foundation Enterprises, Inc. (Other)
Responsible Party: Principal Investigator, Phillip Coffin, MD, MIA, Principal Investigator, San Francisco Department of Public Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01DA022155-01 (NIH); R01DA022155 (NIH); 1R01DA022155-01 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Substance Abuse; HIV Infections
Keywords: Methamphetamine; HIV; MSM; HIV Seronegativity
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirtazapine (Active Comparator): mirtazapine 30 mg daily
  Interventions: Drug: mirtazapine
- Placebo (Placebo Comparator): placebo 30 mg daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: mirtazapine — mirtazapine 30 mg daily for 3 months
  Other Names: Remeron
  Arms: Mirtazapine
Drug: placebo — placebo 30 mg daily for 3 months
  Arms: Placebo

SUMMARY:
Studies demonstrate that methamphetamine (meth) use is associated with high-risk sexual behavior among MSM, putting meth-using MSM at extraordinarily high risk for transmitting or acquiring HIV. This study of intermediate size (60 participants) and length (3 months of follow-up) will assess the efficacy of mirtazapine in reducing methamphetamine use among high-risk MSM.

DETAILED DESCRIPTION:
Methamphetamine use is especially prevalent among men who have sex with men (MSM). Population-based surveys report methamphetamine use rates 20 times higher among MSM compared with the general population. Methamphetamine use is also a driving force in the MSM HIV epidemic: methamphetamine use has been associated with increased number of sexual partners, unprotected sex acts, and sexually transmitted infection (STI) and HIV acquisition. Despite these alarming data, relatively few interventions have been tested among methamphetamine-using MSM, and no studies have tested the efficacy of pharmacologic interventions in reducing methamphetamine use in this population. In parallel with the continued testing of behavioral approaches, we believe the time has come to test pharmacologic interventions to reduce methamphetamine use among MSM. Pharmacologic approaches to treating substance use have been successful in treating nicotine, alcohol, and heroin dependence. No studies have tested a pharmacologic intervention to reduce methamphetamine use among MSM at high risk for HIV acquisition and transmission. A recent pilot study found that mirtazapine, a drug with dual dopaminergic and serotonergic properties, significantly reduced methamphetamine withdrawal symptoms when compared to placebo over a two-week period among Thai men in a drug probation center. Mirtazapine is a commonly used, FDA-approved antidepressant; however, in the Thai study its effects on methamphetamine withdrawal were independent of its effects on depressive symptoms, suggesting a direct effect of mirtazapine on treating methamphetamine dependence. We propose to expand upon these promising pilot results by conducting a study of intermediate size (60 participants) and length (3 months of follow-up) to assess the efficacy of mirtazapine in reducing methamphetamine use among high-risk MSM.

The specific aims of our study are:

1. To test the hypothesis that mirtazapine 30 mg daily will reduce methamphetamine use significantly more than placebo among methamphetamine-dependent MSM, as determined by the proportion of methamphetamine-negative urines and by self-report of methamphetamine use in the mirtazapine versus placebo group.
2. To measure the acceptability of mirtazapine and placebo among methamphetamine-dependent MSM, by determining (via electronic pill caps and self-report) medication adherence to mirtazapine and placebo.
3. To measure the safety and tolerability of mirtazapine and placebo among methamphetamine-dependent MSM, as determined by the number of adverse clinical events in the mirtazapine and placebo arms.

If promising, study results will be used to design a phase III clinical trial to determine if mirtazapine's effects on reducing methamphetamine use lead to reductions in methamphetamine-associated sexual risk. We have chosen first to conduct a 3-year intermediate-sized trial in order to determine if mirtazapine reduces methamphetamine use and whether mirtazapine demonstrates good acceptability and tolerability among a population with methamphetamine-associated high-risk sexual behaviors. If this proves to be the case, we believe our study results will provide strong support for a much larger trial to test the hypothesis that mirtazapine-driven reductions in methamphetamine use will result in corresponding decreases in sexual risk behavior. This study is therefore designed to reflect the structure of a larger HIV-risk reduction trial and includes both substance use and sexual risk behavior measures. We will enroll sexually active, methamphetamine-dependent MSM (either HIV-negative or HIV-positive) who will be randomized 1:1 to receive mirtazapine or placebo for 90 days. Because no medications have been approved to treat methamphetamine dependence, we include extensive safety parameters, as is required by the Food and Drug Administration (FDA) when testing a medication for a new indication in a new population. Participants will be seen weekly for urine drug testing and for brief substance use counseling. All will receive HIV risk-reduction counseling. Behavior will be assessed using standardized measures via audio computer-assisted self-interview (ACASI).

ELIGIBILITY:
Inclusion Criteria:

1. HIV-negative by rapid test, or documentation of HIV infection with a laboratory result of a positive HIV test;
2. male gender;
3. reports having anal sex with men in the prior 3 months while using methamphetamine;
4. diagnosed with methamphetamine dependence as determined by SCID;
5. interested in stopping or reducing methamphetamine use;
6. at least one methamphetamine-positive urine at screening and run-in period;
7. no known allergies to mirtazapine;
8. no current acute illnesses requiring prolonged medical care;
9. no chronic illnesses that are likely to progress clinically during trial participation;
10. able and willing to provide informed consent and to be followed over a 3-month period;
11. age 18-60 years;
12. baseline CBC, total protein, albumin, glucose, alk phos, creatinine, BUN and electrolytes without clinically significant abnormalities as determined by investigator in conjunction with symptoms, physical exam, and medical history.

Exclusion Criteria:

1. evidence of current major depression, as determined by SCID;70
2. history of bipolar disorder or psychosis, as determined by SCID;
3. taking anti-depressant or other psychotropic medication within the last 30 days, including mirtazapine or a monoamine oxidase (MAO) inhibitor;
4. currently using or unwilling not to use pseudoephedrine-containing products for trial duration (causes false positive urines for methamphetamine use);
5. current CD4 count < 200 cells/mm3;
6. measured moderate or severe liver disease (AST, ALT, and total bilirubin > 3 times upper limit of normal) and/or any symptoms of current liver disease;
7. impaired renal function (creatinine clearance < 60 ml/min);
8. currently participating in another research study;
9. any condition that, in the principal investigator's judgment, interferes with safe study participation or adherence to study procedures.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant N Colfax, MD, Principal Investigator — Co-Directior, HIV Epidemiology Section, San Francisco Department of Public Health
Locations (1):
- San Francisco Department of Public Health, Substance Use Research Unit, San Francisco, California, United States

REFERENCES:
- [Result] Colfax GN, Santos GM, Das M, Santos DM, Matheson T, Gasper J, Shoptaw S, Vittinghoff E. Mirtazapine to reduce methamphetamine use: a randomized controlled trial. Arch Gen Psychiatry. 2011 Nov;68(11):1168-75. doi: 10.1001/archgenpsychiatry.2011.124. PMID 22065532

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator:: mirtazapine 30 mg daily for 3 months
- Placebo Comparator:: placebo 30 mg daily for 3 months
Period: Overall Study
Arm/Group | Active Comparator: | Placebo Comparator:
Started | 30 | 30
Completed | 28 | 28
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: | Placebo Comparator: | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (8.0) | 40.1 (10.1) | 40.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 30 | 60
Race/Ethnicity, Customized [Number; unit: participants]
  White | 18 (60) | 19 (63) | 37
  African American | 6 (20) | 5 (17) | 11
  Latino | 3 (10) | 4 (13) | 7
  Other | 3 (10) | 2 (7) | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Positive Methamphetamine Urine Tests, Comparing Baseline (Week 0) to Final Visit (Week 12).
Time Frame: Baseline (week 0) and Final Visit (week 12)
Measure: Number; unit: Percentage reduction
Arm/Group | Active Comparator: | Placebo Comparator:
Number analyzed (Participants) | 30 | 30
Percentage reduction | 40 | 6

2. Primary Outcome: Proportion of Days With Recorded Pill Bottle Opening, as Determined by MEMS.
Description: Proportion of days with recorded pill bottle opening, as determined by MEMS (medication event monitoring system).
Time Frame: Daily, from Baseline (week 0) through Final Visit (week 12)
Measure: Mean (Standard Deviation); unit: Percentage of recorded openings
Arm/Group | Active Comparator: | Placebo Comparator:
Number analyzed (Participants) | 30 | 30
Percentage of recorded openings | 48.3 (26.9) | 48.7 (26.9)

3. Primary Outcome: Frequency of Adverse Events Reported
Time Frame: From Baseline (week 0) through Final Visit (week 12)
Measure: Number; unit: Adverse Events Reported
Arm/Group | Active Comparator: | Placebo Comparator:
Number analyzed (Participants) | 30 | 30
Adverse Events Reported | 109 | 107

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Active Comparator: | Placebo Comparator:
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/30
Other Adverse Events (participants affected / at risk) | 27/30 | 24/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: (N=30) | Placebo Comparator: (N=30)
Compression (spine) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meth-induced Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: (N=30) | Placebo Comparator: (N=30)
Drowsiness (Nervous system disorders) | 13 (19) | 0 (0)
Increased ALT (Hepatobiliary disorders) | 7 (10) | 9 (12)
Increased AST (Hepatobiliary disorders) | 5 (7) | 8 (11)
Gastroenteritis (Gastrointestinal disorders) | 4 (4) | 4 (4)
Gonorrhea (Infections and infestations) | 3 (3) | 1 (1)
Increased Creatinine (Renal and urinary disorders) | 2 (2) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (5) | 3 (4)
Hyperbilirubinemia (Hepatobiliary disorders) | 2 (2) | 4 (5)
Increased Appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Weight Gain (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
Skin and Soft Tissue Infection (Infections and infestations) | 3 (3) | 7 (10)
Increased Alkaline Phosphatase (Hepatobiliary disorders) | 1 (1) | 4 (4)
Insomnia (Nervous system disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No